CLINICAL TRIAL: NCT03219073
Title: Transcranial Direct Current Stimulation to Lower Neuropathic Pain in People With Multiple Sclerosis: a Mechanistic FDG-PET Study
Brief Title: Transcranial Direct Current Stimulation to Lower Neuropathic Pain in People With Multiple Sclerosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator is taking appointment with another institution.
Sponsor: Thorsten Rudroff (Other)
Responsible Party: Sponsor-Investigator, Thorsten Rudroff, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0690
Record Dates: First submitted 2017-04-14; First posted 2017-07-17 (Actual); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis; Neuropathic Pain
Keywords: multiple sclerosis; neuropathic pain; [18F] FDG-PET CT; tDCS; transcranial direct current stimulation
MeSH Terms: conditions — Multiple Sclerosis; Neuralgia

STUDY DESIGN:
Intervention Model Description: Two age and sex matched groups, each n =8, will be randomized to receive either tDCS or SHAM stimulation.
Who Masked: Participant, Care Provider
Masking Description: Patients and assessing investigator will be blinded to group allocation while the treating investigator, who has to set the tDCS or sham-stimulation protocol on the stimulator, will be the only person aware of the stimulation condition. To minimize communication between blinded and non-blinded participants, the treating investigator will be instructed not to talk to patients and the assessing investigator about the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SHAM tDCS (Sham Comparator): SHAM tDCS using tDCS device will be used for sham stimulation where the electrodes will be placed in the same positions as for anodal M1 stimulation, but the stimulator will be turned off after 90 seconds. Therefore, the patients feel the initial itching sensation but receive no current for the rest of the stimulation period.
  Interventions: Device: SHAM tDCS using tDCS device
- Active tDCS with a tDCS device (Active Comparator): Active tDCS using tDCS device (Neuroelectrics Inc., Simi Valley, CA, USA) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The anodal electrode will be placed over the M1 contralateral to the worst somatic pain area (C3, EEG 10/20 system) and the cathode over the supraorbital area contralateral to the anodal electrode. A constant current of 2 mA intensity will be applied for 20 minutes once a day for 5 consecutive days.
  Interventions: Device: Active tDCS using tDCS device

INTERVENTIONS:
Device: Active tDCS using tDCS device — Active tDCS using tDCS device is a noninvasive brain stimulation technique that utilizes low amplitude direct currents applied via scalp electrodes to apply currents to the brain and modulate the level of cortical excitability. tDCS applied over the dorsolateral prefrontal and motor cortex has been reported to be able to decrease pain sensation and to increase pain threshold in healthy subjects and is effective in reducing central chronic pain in PwMS.
  Arms: Active tDCS with a tDCS device
Device: SHAM tDCS using tDCS device — SHAM tDCS emulates active tDCS in all but the actual stimulation. Electrodes of the tDCS device are placed in the same place as with active tDCS however no current is activated.
  Arms: SHAM tDCS

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) is a noninvasive brain stimulation technique that utilizes low amplitude direct currents applied via scalp electrodes to apply currents to the brain and modulate the level of cortical excitability. tDCS applied over the dorsolateral prefrontal and motor cortex has been reported to be able to decrease pain sensation and to increase pain threshold in healthy subjects and is effective in reducing central chronic pain in patients with multiple sclerosis (PwMS.) In spite of the encouraging results of tDCS in PwMS, detailed mechanisms accounting for its analgesic effect have not yet been elucidated.

This will be the first study to determine the effects of tDCS on whole and regional brain activity in PwMS with neuropathic pain to identify potential mechanisms of the analgesic effects of tDCS. These findings will provide targets for future studies investigating different stimulation areas, possible short- and long-term side effects, and specific target areas for other precise stimulation techniques such as transcranial magnetic stimulation.

DETAILED DESCRIPTION:
The investigators aim is to identify changes in brain activation following transcranial direct current stimulation (tDCS), and determine whether these changes are associated with reduced ratings of pain. The investigators hypothesize that the analgesic effects of tDCS are associated with altered glucose metabolism of key regions of the top-down pain modulatory system, such as the dorsolateral prefrontal cortex (DLPFC) and medulla.

This study will follow an interventional protocol with two groups. Upon enrollment into the study, all participants will undergo testing for the outcome measures described above. Each participant will then be randomly assigned into the SHAM or tDCS group for the study intervention. This study will be completed over the course of 6 consecutive days and 1 follow-up phone call 1 week after the final testing for each participant (total of 13 days).

Two age and sex matched groups, each n =8, will receive either tDCS or SHAM stimulation.

All of the following measures will be performed before and after the tDCS or SHAM intervention.

Fluorodeoxyglucose ([18F] FDG) - Whole and regional brain FDG uptake will be measured to determine the mechanistic effect of tDCS on brain activity.

Visual Analog Scale (VAS) - The VAS is a self-evaluation scale where the participant is asked to mark a segment that ranges from 0-100 as visually described in millimeter units where 0 mm indicates no pain and 100 mm indicates the worst possible pain. This scale has been widely used in studies that evaluated pain as an outcome measure: both validity and reproducibility have been demonstrated.

VAS for Anxiety - This is a self-evaluation scale that ranges from 0 to 100 mm: 0 mm indicates no anxiety and 100 mm indicates the worst possible anxiety.

Prior to beginning the 2nd-5th tDCS sessions, the effectiveness of tDCS will be assessed using the following procedures:

Visual Analog Scale (VAS) - Each participant will be asked how effective the previous day's tDCS session was at reducing their pain by marking a segment on the range of 0-100 as visually described in millimeter units where 0 mm indicates no reduction in pain and 100 mm indicates complete alleviation of pain.

Duration of Relief - If the participant indicates any reduction in pain following the previous day's tDCS session, the participant will be asked to estimate how long the participant's pain was reduced following the session.

One week following the post-intervention testing, participants will be contacted via telephone and asked the following questions:

1. Was tDCS effective at reducing the participant's pain?
2. If so, how long did the participant notice a reduction in pain following the participant's final tDCS session?
3. Have the participants reduced their use of pain relieving medications since the last tDCS session?

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple Sclerosis (PwMS)
* Age range 18-65
* Expanded disability status scale comprised between 1.5 and 6.5 with relapsing remitting MS (RRMS) in remitting phase
* Presenting with chronic, drug-resistant, neuropathic pain
* Patients must score at or above a 0 on the Neuropathic Pain Questionnaire (NPQ).
* Patients must score at least a 40 mm on the visual analog scale (VAS) for pain perception at baseline
* All analgesic medications discontinued at least 24 hours before entering the study

Exclusion Criteria:

* Any change in:

  * disease-modifying medications, or
  * a relapse of disease symptoms within the last 60 days
* History of seizures
* History of traumatic brain injury
* History of claustrophobia
* Presence of:

  * pacemakers,
  * aneurysm clips,
  * artificial heart valves,
  * metallic prostheses, or
  * pregnancy.
* Recent hospitalization (within the last 3 months)
* Enforced bed rest/sedentary state
* Resting plasma glucose greater than 200 mg/dl
* Presence of other neurological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Rudroff, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one person completed the the study. Problems with recruitment of more subjects.
Period: Overall Study
Arm/Group | SHAM tDCS | Active tDCS With a tDCS Device
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: For this pilot study we only had one subject who received Active tDCS.
Arm/Group | Active tDCS With a tDCS Device
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Glucose Uptake in Patients With Multiple Sclerosis With Neuropathic Pain
Description: Whole and regional brain glucose uptake via positron emission tomography with a glucose analogue tracer will be measured to determine the mechanistic effect of transcranial direct current stimulation on brain activity in subjects. Glucose uptake will be determined in patients with multiple sclerosis who received brain stimulation and patients with multiple sclerosis who received SHAM. The outcome variable is the mean Standardized Uptake Value.
Time Frame: 1 week
Population: For this pilot study we only had one subject with active transcranial direct current stimulation.
Measure: Mean (Standard Deviation); unit: percentage of glucose uptake increase
Arm/Group | Active tDCS With a tDCS Device
Number analyzed (Participants) | 1
percentage of glucose uptake increase | 3 (0)

2. Secondary Outcome: Change in Neuropathic Pain as Recorded on a Visual Analog Scale (VAS).
Description: VAS Scale 0-100 The higher the worse.
Time Frame: 1 week
Population: For this pilot study we only had one subject with Active tDCS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tDCS With a tDCS Device
Number analyzed (Participants) | 1
units on a scale | 64 (0)

3. Secondary Outcome: Change in Neuropathic Symptom Inventory
Description: The neuropathic symptom inventory is a 12-item questionnaire. This is a valid and reliable measure of neuropathic pain in adults. The Neuropathic Pain Symptoms Inventory (NPSI) contains 12 items in 5 subscales. The subscales include superficial and deep spontaneous pain, paroxysmal pain, evoked pain, and dysesthesia/paresthesia. Among the 12 items, 10 are scored using a numerical rating scale (NRS), ranging from 0 to 10, assessing the severity of experienced neuropathic pain within the previous 24 hours.
  Higher scores of NPSI indicate more severe peripheral neuropathy.10 is the highest score and indicates severe peripheral neuropathy.
  Minimum score is 0 and the maximum score is 120.
Time Frame: 1 week
Population: For this pilot study we only had one subject with active transcranial direct current stimulation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active Transcranial Direct Current Stimulation: Active tDCS using tDCS device (Neuroelectrics Inc., Simi Valley, CA, USA) will deliver a small direct current through two sponge surface electrodes (5cm × 5cm, soaked with 15 mM NaCL). The anodal electrode will be placed over the M1 contralateral to the worst somatic pain area (C3, EEG 10/20 system) and the cathode over the supraorbital area contralateral to the anodal electrode. A constant current of 2 mA intensity will be applied for 20 minutes once a day for 5 consecutive days.
  Active tDCS using tDCS device: Active tDCS using tDCS device is a noninvasive brain stimulation technique that utilizes low amplitude direct currents applied via scalp electrodes to apply currents to the brain and modulate the level of cortical excitability. tDCS applied over the dorsolateral prefrontal and motor cortex has been reported to be able to decrease pain sensation and to increase pain threshold in healthy subjects and is effective in reducing central chronic pain in PwMS.
Arm/Group | Active Transcranial Direct Current Stimulation
Number analyzed (Participants) | 1
units on a scale | 68 (0)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Active tDCS With a tDCS Device
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03219073/Prot_005.pdf